CLINICAL TRIAL: NCT03495089
Title: Feasibility and Effectiveness of Electrochemical Dermal Conductance Measurement for the Screening of Diabetic Neuropathy in Primary Care.
Brief Title: DECODING Study (Dermal Electrochemical Conductance in Diabetic Neuropathy)
Acronym: DECODING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: P14/147
Record Dates: First submitted 2018-03-19; First posted 2018-04-11 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-04

CONDITIONS: Neuropathy, Diabetic; Diabetes Mellitus, Type 2
Keywords: Screening; Sudomotor reflex; DEC; Primary Care
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2; Hamartoma Syndrome, Multiple

STUDY DESIGN:
Intervention Model Description: consecutively there will be included patients with type 2 DM over 40 years of age, with or without symptoms of neuropathy, attended in Primary Care. We will also include the following two groups of patients matched by age and gender: one including patients with prediabetes (intermediate alterations of glucose metabolism defined as impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) determined by OGTT after 2-hour 75 g oral glucose administration and another including patients without glucose alterations (normal glucose tolerance) (control group)
Who Masked: Investigator
Masking Description: A neurologist will be blinded to previous test results and will perform neurographyc test including sensory conduction study of the median, ulnar and sural nerves, and motor conduction study of the deep peroneal nerve.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with type 2 DM (Experimental): Patients with type 2 DM over 40 years of age, with or without symptoms of neuropathy, attended in Primary Care.
  Intervention(s) to be administered:After verifying the inclusion criteria and receiving written informed consent to participate, during the first visit to the Primary Care centres the medical history of the patient will be obtained and a physical examination will be performed using the Monofilament testing -MFT and the Neuropathy Disability Score-NDS and Utah Early Neuropathy Scale-UENS questionnaires will be given to screen for polyneuropathy-PN. The patient will also undergo dermal electrochemical conductance- DEC quantification using the Sudoscan® device.
  Interventions: Diagnostic Test: dermal electrochemical conductance (DEC); Diagnostic Test: Monofilament testing
- prediabetes (Experimental): Patients with intermediate alterations of glucose metabolism defined as impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) determined by OGTT after 2-hour 75 g oral glucose administration.
  Intervention(s) to be administered:After verifying the inclusion criteria and receiving written informed consent to participate, during the first visit to the Primary Care centres the medical history of the patient will be obtained and a physical examination will be performed using the Monofilament testing -MFT and the Neuropathy Disability Score-NDS and Utah Early Neuropathy Scale-UENS questionnaires will be given to screen for polyneuropathy-PN. The patient will also undergo dermal electrochemical conductance-DEC quantification using the Sudoscan® device.
  Interventions: Diagnostic Test: dermal electrochemical conductance (DEC); Diagnostic Test: Monofilament testing
- control group (Experimental): Patients without glucose alterations (normal glucose tolerance). Intervention(s) to be administered:After verifying the inclusion criteria and receiving written informed consent to participate, during the first visit to the Primary Care centres the medical history of the patient will be obtained and a physical examination will be performed using the Monofilament testing -MFT and the Neuropathy Disability Score-NDS and Utah Early Neuropathy Scale-UENS questionnaires will be given to screen for polyneuropathy-PN. The patient will also undergo dermal electrochemical conductance-DEC quantification using the Sudoscan® device.
  Interventions: Diagnostic Test: dermal electrochemical conductance (DEC); Diagnostic Test: Monofilament testing

INTERVENTIONS:
Diagnostic Test: dermal electrochemical conductance (DEC) — The patient will undergo DEC quantification using the Sudoscan® device.(Sudoscan®, Impeto Medical, France)
Diagnostic Test: Monofilament testing — Monofilament testing by Semmes-Weinstein 5:07 MFT (10 g),

SUMMARY:
Diabetes mellitus is the leading cause of polyneuropathy in the Western world. Diabetic neuropathy is a frequent complication of diabetes and may have great clinical transcendence due to pain and possible ulceration of the lower extremities. It is also a relevant cause of morbidity and mortality in patients with diabetes. Although the cause of polyneuropathy in patients with diabetes is only partially known, it has been associated with chronic hyperglycaemia suggesting the possible aetiopathogenic implication of advanced glycosylation end-products. The strategy of choice in the medical management of diabetic neuropathy is early detection since glycaemic control and the use of certain drugs may prevent or slow the development of this disease. Diabetic neuropathy most often presents with a dysfunction of unmyelinated C-fibers, manifested as an alteration of the sweat reflex of the eccrine glands. This dysfunction can now be demonstrated using a newly developed technology which measures dermal electrochemical conductivity. This noninvasive test is easy and cost-effective. The aim of the present study is to evaluate the feasibility and effectiveness of dermal electrochemical conductance measurement (quantitative expression of the sudomotor reflex) as a screening test for the diagnosis of diabetic neuropathy in patients in primary care.

DETAILED DESCRIPTION:
The prevalence of diabetes mellitus (DM) is very high in Spain, being nearly 14% according to oral glucose tolerance test (OGTT) results . The management of DM requires a significant consumption of healthcare resources, mainly in relation to the care of vascular complications. Among the late microvascular events which may develop in patients with DM, polyneuropathy (PN) is the most common and disabling, and is the leading cause of morbidity and mortality in these patients. Indeed, in Spain, the leading cause of neuropathy is DM, with its prevalence increasing with the presence of DM and other risk factors such as obesity.

PN is defined as the presence of symptoms and/or signs of peripheral nerve dysfunction in people with DM after the exclusion of other possible causes. The Toronto Panel Consensus on PN defined this disorder as "symmetrical, depending on large fibers, sensory-motor attributable to metabolic and micro vessel disorders, as a result of chronic hyperglycemia and other risk factors". In patients with PN, thin fibers (autonomic system - sweating) and thermal and tactile sensitivity are first affected, followed by the involvement of large fibers, presenting an altered vibrating sensation which eventually alters electromyography (EMG) patterns. Therefore, dysfunction of sweat reflex in small distal fibers is one of the earliest changes to be detected in these patients.

The most common clinical presentation of PN is distal symmetric polyneuropathy (DSPN), being predominantly sensory in 80% of cases. Pain is the most important symptom, being described as burning or flashing, lancinating, deep, and with frequent exacerbations during rest (4). Pain often affects the quality of life of these patients, and it is a frequent cause of depression and/or anxiety. Moreover, some patients may develop hypoesthesia, which may lead to severe foot lesions.

The prevalence of DSPN varies greatly according to the population, definition and detection method. The Rochester study, including more than 64,000 patients, reported the prevalence of PN to be between 66% and 59% for type1 DM and type 2 DM, respectively. The 3rd report of the Technical Study Group of Diabetes of the World Health Organization (WHO) described a prevalence of 40% (8), and 50% in patients with more than 25 years of DM evolution. Pirart et al. reported a prevalence ranging from 25 to 48% (7,10-17), while in Spain, Cabezas-Cerrato et al. published a figure of 24.1%. DSPN-related factors are: age, DM duration, metabolic control, male gender, acute myocardial infarction, hyperlipidemia (especially hypertriglyceridemia), smoking, and general cardiovascular risk factors . Puig et al. also included urinary albumin excretion as a risk factor of presenting DSPN.

The diagnosis of DSPN is commonly made based on signs and symptoms and usually includes the use of several questionnaires such as the Neuropathy Disability Score (NDS), the Neuropathy Symptoms Score (NSS) and the Michigan Neuropathy Instrument (MNI). These questionnaires are easy to perform and are reproducible, sensitive and adequate for use in a screening program. Additionally, It was included a short scale (UENS - Utah Early Neuropathy Scale) to screen early neuropathy . This sensitive, fast and practical test, has 5 items and their score ranges from 0 to 42 points.

There are many confirmatory tests, including measurements of nerve conduction velocity (EMG) and bio-thesiometry or skin biopsy. However, those most commonly used are the measurement of altered sensations using a vibrating tuning fork with 128 Hz and/or pressure with Semmes-Weinstein 5:07 monofilament. Monofilament testing (MFT) is widely accepted and recommended by all scientific societies because of its validity, predictive risk, efficiency and simplicity. Feng et al. reported that MFT has a sensitivity of 57-93%, a specificity of 75-100%, a positive predictive value of 36-94% and a negative predictive value of 84-100% compared to the measurement of nerve velocity by EMG. Although electrophysiological measures are more objective and reproducible, they are limited in that they only detect dysfunction based on the presence of thicker and faster (myelinated) fibers and show their involvement later. Consequently, EMG is a specific, albeit very insensitive, test.

Recently developed noninvasive techniques are more reproducible and reliable for the detection of early dysfunction of small fibers. One of these new techniques involves the measurement of dermal electrochemical conductance (DEC) or sudomotor dysfunction index and has been evaluated by well-designed studies (Calvet, Dupin, Winiecki, Black, 2013; Casellini 2013; Devigili 2008; Peltier 2009) which support its use as a screening test .

Ramachandran et al studied the use of DEC to detect diabetes and other disorders of glucose metabolism. In a study on the use of DEC Casellini et al (5) applied a PN test which showed a low sensitivity of 78% and a specificity of 92% in diabetic patients without neuropathy compared to other subjects with neuropathy and a control group. In this latter study, correlation with clinical parameters showed adequate reproducibility of the results, particularly in regard to the measurements of the feet . Several other studies also obtained significantly lower DEC values on comparing diabetic patients and controls. In a study of patients following a 12-month program of intense physical activity, Raisanen et al (23) observed a greater improvement in DEC compared to weight, waist circumference or maximum oxygen volume (VO2 max).

Therefore, taking into account the large number of methods used and the learning curve required to correctly implement these techniques as well as the absence of consensus as to which method is the most adequate to diagnose DSPN, the aim of this study is to validate the usefulness of DEC measurement in the early diagnosis of DSPN compared with traditional techniques in the Primary Care setting.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 DM
* patients with pre-diabetes
* patients without glucose alterations

Three main diagnostic categories (normal, pre-diabetes and diabetes) were defined using the WHO criteria based on 2-h postload glucose [<7.8 (140 mg/dL), 7.8-11.0 mmol/L (140-200 mg/dL) and / or fasting plasma glucose (6.1-6.9 mmol/L; 110-126 mg/dL) and >11.1 mmol/L (>200 mg/dL), respectively.

Exclusion Criteria:

* Type 1 DM
* upper or lower limb amputation (except phalanges),
* diagnosis of neuropathy not related to diabetes
* neuropathy by entrapment
* use of psychoactive substances
* chronic alcoholism
* malnutrition
* treatment with beta-blockers
* presence of terminal disease or life expectancy less than 3 years

Pregnancy will be ruled out in women (negative pregnancy test) and a possible history of gestational diabetes will also be taken into account.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Presence of diabetic neuropathy diagnosed by EMG | Day 1
  Presence of diabetic neuropathy diagnosed by electromyography

SECONDARY OUTCOMES:
Neuropathy Disability Score | Day 1
  Presence of diabetic neuropathy diagnosed by Neuropathy Disability Score (NDS). - A NDS score greater than or equal to 6 points will be considered as the presence of diabetic neuropathy.
Utah Early Neuropathy Scale | Day 1
  Presence of diabetic neuropathy diagnosed by Utah Early Neuropathy Scale (UENS). A UENS score greater than or equal to 10 points will be considered as the presence of diabetic neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Costa, MD, Study Chair — Jordi Gol Primary Care Research Institute, Catalan Health Institute, Primary Health Care Division, Reus-Barcelona, Catalonia, Spain
Locations (3):
- Spain (3):
  - Hospital Universitari Mútua Terrassa, Terrassa, Barcelona
  - Mútua Terrassa Primary Care, Terrassa, Barcelona
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Soriguer F, Goday A, Bosch-Comas A, Bordiu E, Calle-Pascual A, Carmena R, Casamitjana R, Castano L, Castell C, Catala M, Delgado E, Franch J, Gaztambide S, Girbes J, Gomis R, Gutierrez G, Lopez-Alba A, Martinez-Larrad MT, Menendez E, Mora-Peces I, Ortega E, Pascual-Manich G, Rojo-Martinez G, Serrano-Rios M, Valdes S, Vazquez JA, Vendrell J. Prevalence of diabetes mellitus and impaired glucose regulation in Spain: the Di@bet.es Study. Diabetologia. 2012 Jan;55(1):88-93. doi: 10.1007/s00125-011-2336-9. Epub 2011 Oct 11. PMID 21987347
- [Background] Tesfaye S, Selvarajah D. Advances in the epidemiology, pathogenesis and management of diabetic peripheral neuropathy. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:8-14. doi: 10.1002/dmrr.2239. PMID 22271716
- [Background] Said G. Diabetic neuropathy--a review. Nat Clin Pract Neurol. 2007 Jun;3(6):331-40. doi: 10.1038/ncpneuro0504. PMID 17549059
- [Background] Samper Bernal D, Monerris Tabasco MM, Homs Riera M, Soler Pedrola M. Etiología y manejo de la neuropatía diabética dolorosa. Rev Soc Esp Dolor. 2010;17(6):286-96. [article in Spanish].
- [Background] Casellini CM, Parson HK, Richardson MS, Nevoret ML, Vinik AI. Sudoscan, a noninvasive tool for detecting diabetic small fiber neuropathy and autonomic dysfunction. Diabetes Technol Ther. 2013 Nov;15(11):948-53. doi: 10.1089/dia.2013.0129. Epub 2013 Jul 27. PMID 23889506
- [Background] Gore M, Brandenburg NA, Dukes E, Hoffman DL, Tai KS, Stacey B. Pain severity in diabetic peripheral neuropathy is associated with patient functioning, symptom levels of anxiety and depression, and sleep. J Pain Symptom Manage. 2005 Oct;30(4):374-85. doi: 10.1016/j.jpainsymman.2005.04.009. PMID 16256902
- [Background] Tesfaye S, Stevens LK, Stephenson JM, Fuller JH, Plater M, Ionescu-Tirgoviste C, Nuber A, Pozza G, Ward JD. Prevalence of diabetic peripheral neuropathy and its relation to glycaemic control and potential risk factors: the EURODIAB IDDM Complications Study. Diabetologia. 1996 Nov;39(11):1377-84. doi: 10.1007/s001250050586. PMID 8933008
- [Background] Vidal MA, Martínez-Fernández E, Martínez-Vázquez de Castro J, Torres LM. Neuropatía diabética. Eficacia de la amitriptilina y de la gabapentina. Rev Soc Esp Dolor. 2004;11:490-504 [article in Spanish].
- [Background] Pirart J. Diabetes mellitus and its degenerative complications: a prospective study of 4,400 patients observed between 1947 and 1973. Diabetes Care. 1978;1(3):168-88.
- [Background] Dyck PJ, Kratz KM, Karnes JL, Litchy WJ, Klein R, Pach JM, Wilson DM, O'Brien PC, Melton LJ 3rd, Service FJ. The prevalence by staged severity of various types of diabetic neuropathy, retinopathy, and nephropathy in a population-based cohort: the Rochester Diabetic Neuropathy Study. Neurology. 1993 Apr;43(4):817-24. doi: 10.1212/wnl.43.4.817. PMID 8469345
- [Background] Cabezas-Cerrato J. The prevalence of clinical diabetic polyneuropathy in Spain: a study in primary care and hospital clinic groups. Neuropathy Spanish Study Group of the Spanish Diabetes Society (SDS). Diabetologia. 1998 Nov;41(11):1263-9. doi: 10.1007/s001250051063. PMID 9833931
- [Background] Gómez MA GM. Estudio de la conduccion nerviosa en pacientes con diabetes mellitus tipo 2. Rev Peru Endocrinol Metab. 1998;IV:23-33. [article in Spanish].
- [Background] Lu B, Hu J, Wen J, Zhang Z, Zhou L, Li Y, Hu R. Determination of peripheral neuropathy prevalence and associated factors in Chinese subjects with diabetes and pre-diabetes - ShangHai Diabetic neuRopathy Epidemiology and Molecular Genetics Study (SH-DREAMS). PLoS One. 2013 Apr 16;8(4):e61053. doi: 10.1371/journal.pone.0061053. Print 2013. PMID 23613782
- [Background] Ziegler D, Papanas N, Rathmann W, Heier M, Scheer M, Meisinger C; KORA Study Group. Evaluation of the Neuropad sudomotor function test as a screening tool for polyneuropathy in the elderly population with diabetes and pre-diabetes: the KORA F4 survey. Diabetes Metab Res Rev. 2012 Nov;28(8):692-7. doi: 10.1002/dmrr.2340. PMID 22949335
- [Background] Puig ML, Aguirre DR, Rodríguez MC, Alonso ED. Neuropatía periférica de los miembros inferiores en diabéticos tipo 2 de diagnóstico reciente. Av Endocrinol 2006;22(2):149. [article in Spanish].
- [Background] Calle Pascual AL, Runkle Vega I, Díaz Pérez JA, Durán Hervada A, Romero Pérez L. Técnicas de exploración. Av Diabetol. 2006;22(1):42-9. [article in Spanish].
- [Background] Singleton JR, Bixby B, Russell JW, Feldman EL, Peltier A, Goldstein J, Howard J, Smith AG. The Utah Early Neuropathy Scale: a sensitive clinical scale for early sensory predominant neuropathy. J Peripher Nerv Syst. 2008 Sep;13(3):218-27. doi: 10.1111/j.1529-8027.2008.00180.x. PMID 18844788
- [Background] Kanji JN, Anglin RE, Hunt DL, Panju A. Does this patient with diabetes have large-fiber peripheral neuropathy? JAMA. 2010 Apr 21;303(15):1526-32. doi: 10.1001/jama.2010.428. PMID 20407062
- [Background] Feng Y, Schlosser FJ, Sumpio BE. The Semmes Weinstein monofilament examination as a screening tool for diabetic peripheral neuropathy. J Vasc Surg. 2009 Sep;50(3):675-82, 682.e1. doi: 10.1016/j.jvs.2009.05.017. Epub 2009 Jul 30. PMID 19595541
- [Background] Smith AG, Lessard M, Reyna S, Doudova M, Singleton JR. The diagnostic utility of Sudoscan for distal symmetric peripheral neuropathy. J Diabetes Complications. 2014 Jul-Aug;28(4):511-6. doi: 10.1016/j.jdiacomp.2014.02.013. Epub 2014 Mar 6. PMID 24661818
- [Background] Ramachandran A, Moses A, Shetty S, Thirupurasundari CJ, Seeli AC, Snehalatha C, Singvi S, Deslypere JP. A new non-invasive technology to screen for dysglycaemia including diabetes. Diabetes Res Clin Pract. 2010 Jun;88(3):302-6. doi: 10.1016/j.diabres.2010.01.023. Epub 2010 Feb 25. PMID 20188429
- [Background] Mayaudon H, Miloche PO, Bauduceau B. A new simple method for assessing sudomotor function: relevance in type 2 diabetes. Diabetes Metab. 2010 Dec;36(6 Pt 1):450-4. doi: 10.1016/j.diabet.2010.05.004. Epub 2010 Aug 23. PMID 20739207
- [Background] Raisanen A, Eklund J, Calvet JH, Tuomilehto J. Sudomotor function as a tool for cardiorespiratory fitness level evaluation: comparison with maximal exercise capacity. Int J Environ Res Public Health. 2014 May 30;11(6):5839-48. doi: 10.3390/ijerph110605839. PMID 24886754
- [Background] Veresiu AI, Bondor CI, Florea B, Vinik EJ, Vinik AI, Gavan NA. Detection of undisclosed neuropathy and assessment of its impact on quality of life: a survey in 25,000 Romanian patients with diabetes. J Diabetes Complications. 2015 Jul;29(5):644-9. doi: 10.1016/j.jdiacomp.2015.04.001. Epub 2015 Apr 9. PMID 25922309

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03495089/Prot_SAP_000.pdf